CLINICAL TRIAL: NCT03981068
Title: DAHANCA 37 A Phase II Study of Intensity Modulated Proton Therapy (IMPT) for Re-irradiation With Curative Intent for Recurrent or New Primary Head and Neck Cancer
Brief Title: DAHANCA 37. Re-irradiation With Proton Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dahanca 37
Record Dates: First submitted 2019-05-30; First posted 2019-06-10 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Neoplasms
Keywords: recurrent; reirradiation; second primary
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — Re-Irradiation; Cisplatin; Nimorazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Re-Irradiation with protons (Experimental): 60 Gy in 50 fraktions, 10 weekly with protons
  Interventions: Radiation: Re-irradiation

INTERVENTIONS:
Radiation: Re-irradiation — Cisplatin for all eligible patients, nimorazole for all SCC
  Other Names: cisplatin; nimorazole

SUMMARY:
Summary Design Phase II observational

Treatment

* 60 Gy/50 fx / 10W-1 at 1.2 Gy/fx

  o i.e. EQD2 tumor=56 Gy, EQD2 late=50.4 Gy at α/β= 10 and 3, respectively
* Proton radiotherapy
* Concomitant cisplatin for eligible patients*
* Nimorazole recommended for SCC* *The concurrent medical treatment (weekly cisplatin and nimorazole) are prescribed according to the national treatment guidelines, and are not part of the experimental treatment.

Endpoints

* Primary:

  o Any new late toxicity grade >=3 according to CTC AE 5.0
* Secondary

  * Side effects according to DAHANCA scoring system
  * Quality of life and PROM according to EORTC C30 and HN43
  * Loco-regional control (LRC)
  * Overall survival (OS)

DETAILED DESCRIPTION:
Summary Design Phase II observational Inclusion criteria

* Histological verified loco-regional recurrence or new primary
* Available dose plan from primary radiotherapy course
* Comparative dose plan with advantages for proton radiotherapy e.g. integral dose
* Dmax dose (0.03 cm3) on the cumulated photon dose plan≥90 Gy
* Complete Response (CR)* after initial therapy, except in the case where the recurrence is considered a geometric miss (recurrence center of mass (COM) outside the 95% of prescription dose.
* Inoperable or salvage surgery with R1/R2 resection, extranodal extension (ENE) or extensive soft tissue infiltration
* Absence of distant metastasis at both

  * clinical examination AND
  * PET-CT or CT of thorax and upper abdomen
* Life expectancy due to age and co-morbidity of >=1 year. The general condition must be sufficient to tolerate persistent significant side effects, e.g. tube or cannulae
* PS<=2 (WHO See appendix)
* The patients should be able to read Danish in order to participate with quality of life questionnaires, but can participate in the rest of the protocol without being fluent in Danish, if capable of reading the patient information.

  * Complete Response is defined as the situation when a trained clinician, ideally at a multidisciplinary team conference, defines the patient as in complete remission, based on clinical examination and available imaging. This status can of course later be considered wrong as new information becomes available (sub-centimeter nodes grow etc.) Exclusion criteria
* Radical surgery (R0) and absence of adverse prognostic pathological features
* Lymphoma or malignant melanoma
* Inability to attend full course of radiotherapy or follow-up visits in the outpatient clinic
* As of 2019, patients with tracheal cannulas are excluded due to dose uncertainties. This may change if a technical solution becomes available.

Treatment

* 60 Gy/50 fx / 10W-1 at 1.2 Gy/fx

  o i.e. EQD2 tumor=56 Gy, EQD2 late=50.4 Gy at α/β= 10 and 3, respectively
* Proton radiotherapy
* Concomitant cisplatin for eligible patients*
* Nimorazole recommended for SCC* *The concurrent medical treatment (weekly cisplatin and nimorazole) are prescribed according to the national treatment guidelines, and are not part of the experimental treatment.

Endpoints

* Primary:

  o Any new late toxicity grade >=3 according to CTC AE 5.0
* Secondary

  * Side effects according to DAHANCA scoring system
  * Quality of life and PROM according to EORTC C30 and HN43
  * Loco-regional control (LRC)
  * Overall survival (OS)

Derived projects

* Morbidity (NTCP) modeling for cumulative doses
* Metrics for uncertainties regarding cumulative doses

ELIGIBILITY:
Inclusion Criteria:

* Histological verified loco-regional recurrence or new primary
* Available dose plan from primary radiotherapy course
* Comparative dose plan with advantages for proton radiotherapy e.g. integral dose
* Dmax dose (0.03 cm3) on the cumulated photon dose plan≥90 Gy
* Complete Response (CR)* after initial therapy, except in the case where the recurrence is considered a geometric miss (recurrence center of mass (COM) outside the 95% of prescription dose.
* Inoperable or salvage surgery with R1/R2 resection, extranodal extension (ENE) or extensive soft tissue infiltration
* Absence of distant metastasis at both

  * clinical examination AND
  * PET-CT or CT of thorax and upper abdomen
* Life expectancy due to age and co-morbidity of >=1 year. The general condition must be sufficient to tolerate persistent significant side effects, e.g. tube or cannulae
* PS<=2 (WHO See appendix)

Exclusion Criteria:

* Radical surgery (R0) and absence of adverse prognostic pathological features
* Lymphoma or malignant melanoma
* Inability to attend full course of radiotherapy or follow-up visits in the outpatient clinic
* As of 2019, patients with tracheal cannulas are excluded due to dose uncertainties. This may change if a technical solution becomes available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Any new grade >=3 toxicity | 3 years after radiotherapy
  CTC AE 5.0

SECONDARY OUTCOMES:
Side effects, any grade | 5 years after radiotherapy
  According to CTC AE or Dahanca
Quality of life and PROM | 6 months
  EORTC QLQ HN43 , swallowing scale. Difference (mean) between baseline and 6 months
Loco-regional control (LRC) | 5 years after radiotherapy -actuarial analysis
  Abscence of locoregional failure
Overall survival (OS) | Median Survival up to 5 years
  Abscence of death

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jensen, Principal Investigator — Danish Centre for Particle Therapy
Locations (1):
- Danish Center for Particle Therapy, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No